CLINICAL TRIAL: NCT03152305
Title: Measure of Intracranial Pressure Variations During Migraine Attacks
Brief Title: Intracranial Pressure During Migraine
Acronym: MigICP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-331; 2014-A00042-45 (Other: 2014-A00042-45)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Menstrual Migraine
Keywords: Migraine; Intracranial pressure; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with menstrual migraine: Womens presenting with regular menstrual migraine treated with triptans will be included in the study.
  Interventions: Other: Intracranial pressure variations
- Matched control: The potential variations will be compared to the measures done on matched healthy women outside and during menses.
  Interventions: Other: Intracranial pressure variations

INTERVENTIONS:
Other: Intracranial pressure variations — Self-measure of ICP will be performed outside and during menstrual migraine attacks.

SUMMARY:
An increase in intracranial pressure (ICP) during migraine attacks is possible and could contribute to pain initiation and maintenance. From now on, it was not possible to measure ICP in a non-invasive way. The development of a new tool allows non-invasive self-measures of ICP variations. Thus, it is possible for the first time to look for such ICP variations during migraine attacks and to conclude if this mechanism is implied in the pathophysiology of migraine.

DETAILED DESCRIPTION:
Womens presenting with regular menstrual migraine treated with triptans will be included in the study. Self-measure of ICP will be performed outside and during menstrual migraine attacks. The potential variations will be compared to the measures done on matched healthy women outside and during menses.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 non menopausal women
* Menstrual migraine
* Using a triptan as usual treatment to relieve attacks
* Usual triptan efficacy although recurrence is possible

Exclusion Criteria:

* Disease of the ear
* Intracranial hypertension
* Chronic daily headache
* Use of topiramate or acetazolamide
* Triptans used more than 10 days/month
* Analgesic drug used more than 15 days/month
* Uncontrolled high blood pressure
* BMI >30
* Ongoing allergic rhinitis or flu

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Womens presenting with regular menstrual migraine treated with triptans will be included in the study. Self-measure of ICP will be performed outside and during menstrual migraine attacks. The potential variations will be compared to the measures done on matched healthy women outside and during menses.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-07-21 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Intracranial pressure variations | during menstrual migraine attacks
  Measured during menstrual migraine attacks compared to ICP in non-migraine days and in matched healthy women

SECONDARY OUTCOMES:
Relationships between ICP variations and clinical parameters | during menstrual migraine attacks
  Age, BMI, pain intensity, pulsating pain, allodynia, nausea, photophobia, phonophobia, dizziness, tinnitus
Relationships between ICP variations and pain relief | during menstrual migraine attacks

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France